CLINICAL TRIAL: NCT01938677
Title: Gamma Knife Radiosurgery vs Initial Conservative Treatment for Vestibular Schwannoma Patients With Preserved Hearing, a Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Petter Forander, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/211-31/1
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Vestibular Schwannoma
Keywords: Vestibular schwannoma; Gamma knife radiosurgery; Hearing preservation
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Gamma knife (Experimental): Patients with VS and preserved hearing, randomized to initial gamma knife radiosurgery will receive this treatment within a few months after enrollment
  Interventions: Radiation: Initial Gamma knife radiosurgery
- Initial conservative (No Intervention): Patients with VS and preserved hearing, randomized to initial conservative treatment will initially be followed with repeated MRI and audiometry. If MRI show progression of VS requiring intervention, patients will receive treatment but still belong to the initial treatment arm, according to intention to treat.

INTERVENTIONS:
Radiation: Initial Gamma knife radiosurgery
  Arms: Initial Gamma knife

SUMMARY:
The effect of Gamma knife radiosurgery (GKRS) on hearing loss, in patients with vestibular schwannoma (VS) and preserved hearing is still unclear. Retrospective data indicate that the hearing is preserved in most patient years after the gamma knife treatment. Recent prospective data suggests that radiosurgery could be a hearing preserving treatment for these patients.

The main objective of this study is to evaluate if GKRS can inhibit progression of hearing loss in patients with VS. Patients with preserved hearing will be offered to participate in the study and randomized ether to GKRS or initial conservative treatment for their vestibular schwannoma. They will then be followed with scheduled magnetic resonance image(MRI) and audiometry and evaluated after one, three and five years after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly (<6 months) diagnosed with Vestibular schwannoma less than 20 mm in diameter.
2. Vestibular schwannoma with or without evidence of growth.
3. Patients between 18 and 80 years of age.
4. Karnofsky performance score >70
5. Patients with vestibular schwannoma and preserved hearing according to Gardner Robertson class 1-2, and speech discrimination (SD) scores between 50-100% will participate in the hearing preservation part of the study.

   -

Exclusion Criteria:

* 1. Patients with Neurofibromatosis type 2 will be excluded to achieve a homogenous study population.

  2. Patients who had other treatments prior to the GKRS (usually microsurgery (MS), GKRS or external beam radiation) for their tumour will also be excluded for the same reason.

  3. Patients who are not citizens in the country where they will be followed will be excluded, to reassure the same follow up within the study population.

  4. Hearing loss due injury or to active ear disease, such as Meniere´s disease, otosclerosis or chronic otitis media.

  5. Patients with poor comprehension of the the language in the country where they are followed, such that adequate performance on speech tests, are unlikely.

  6. Claustrophobia, making MR follow up impossible without sedation. 7. Alcohol- or narcotic abuses that effect compliance to the follow up. 8. Uncontrolled neoplastic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-04; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
The numbers of participants with preserve hearing | up to five years after enrollment
  Baseline audiometric investigation will be performed at time of enrollment. Patients will be followed with audiometric investigations after 1, 3 and 5 years after gamma knife or conservative treatment.Primary endpoint will be numbers of patients with preserve hearing for each treatment arm.

SECONDARY OUTCOMES:
Tumor control | 1, 2, 5 years after enrollment
  MR investigation including digitalized volumetric of vestibular schwannomas will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Karolinska univeristy hospital, Stockholm, Sweden